CLINICAL TRIAL: NCT06985979
Title: Exploring the Needs of High-intensity User Patients Within the Emergency Department: Informing the Development of a Psychosocial Service
Brief Title: Exploring the Needs of HIU Patients Within the Emergency Department
Acronym: HIU ED
Status: Completed | Type: Observational
Sponsor: East Lancashire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: EastLancashireNHS
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: High Intensity Users; Frequent Attenders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Intensity User Patients: Patients who have attended the Emergency Department 5 times or more in the last 12 months.
- Emergency Department Staff: Staff who work in the Emergency Department at Blackburn Royal Teaching Hospital

SUMMARY:
The aim of this qualitative interview study is to explore the unmet needs of patients who frequently attend the emergency department and the challenges of the staff who support them.

The study will interview 10 patients who frequently attend the emergency department and 10 staff members working within the emergency department.

ELIGIBILITY:
Inclusion Criteria:

Patients who have attended the Emergency Department at Blackburn Royal Teaching Hospital over 5 times in the last 12 months All MDT staff within the Emergency Department at Blackburn Royal Teaching Hospital

Exclusion Criteria: Patients under 18 Patients who have not attended the Emergency Department 5 times or more Staff who do not work in the Emergency Department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants of this study will include patients who have been identified by the ED Cerna database to have attended the Emergency Department at Blackburn Royal Teaching Hospital over 5 times in the last 12 months.
  All MDT staff within the Emergency Department at Blackburn Royal Teaching Hospital will be invited to participate (e.g. ED consultants, doctors, junior doctors, nurses as well as reception and portering staff).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Qualitative Interview Data | 2 months
  Qualitative data will be analysed using Reflective Thematic Analysis from telephone interview transcripts.

CONTACTS AND LOCATIONS:
Locations (1):
- Blackburn Royal Teaching Hospital, Blackburn, United Kingdom

IPD SHARING:
Plan to Share IPD: No
I am the only researcher working on this project.